CLINICAL TRIAL: NCT06292026
Title: A Controlled Data Collection and Prospective Treatment Study to Evaluate the Efficacy of ProgenaMatrix™ in the Management of Diabetic Foot Ulcers
Brief Title: Efficacy of ProgenaMatrix™ in the Management of DFUs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProgenaCare Global, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFU/1
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care; Bisphenol A-Glycidyl Methacrylate

STUDY DESIGN:
Intervention Model Description: The objective of this data collection is to look at outcomes and time points for ProgenaMatrix™ in the treatment of diabetic foot ulcers. Additionally, use the collected data to develop predictive wound closure models. There is a 1-week lead in period after initial debridement. If the wound is rapidly moving to closure after initial debridement and standard moist dressings, the withdrawal of these patients will prevent corruption of the true closure rate of ProgenaMatrix™. The objective of the treatment with ProgenaMatrix™ is to evaluate the closure rate in patients not responding to traditional moist therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with ProgenaMatrix (Experimental): application of ProgenaMatrix daily for 12 weeks
  Interventions: Device: ProgenaMatrix Keratin graft; Other: standard of care

INTERVENTIONS:
Device: ProgenaMatrix Keratin graft — place ProgenaMatrix graft on the wound
Other: standard of care — apply non adherent dressing
  Other Names: adaptic

SUMMARY:
This multicenter study will collect data to determine closure time for diabetic ulcers when following protocol parameters and treatment with ProgenaMatrix™.

DETAILED DESCRIPTION:
This is a multicenter data collection and treatment study with weekly updates to include pre and post debridement measurements of wound area, photographs and additional comments of wound appearance, exudate, and patient compliance. ProgenaMatrix™ will be used as the dressing to maintain a moist wound environment post-debridement. ProgenaMatrix™ is US Food and Drug Administration (FDA) cleared for the treatment of diabetic foot ulcers. The standard of care for diabetic foot ulcers (DFU) is removal of non-viable tissue, control of infection, maintain a moist wound environment and off-load the ulcer site. All aspects of this research are within the standard of care practice for the treatment of diabetic foot ulcers.

The use of ProgenaMatrix™ instead of a traditional dressing to maintain a moist healing wound environment is the only research intervention. Data on any adverse events related to treatment with ProgenaMatrix™ will be collected for research purposes.

The data in this study will be collected from subjects with controlled eligibility. The rationale for this control is to provide a real-world data set on subjects that have had their controllable comorbidities attenuated. This is good clinical practice at advanced wound treatment centers. This data will be statistically evaluated to provide a true closure rate when using ProgenaMatrix™ in a subject where standard of care treatments and assessments are followed. As with any good data set the control of as many variables as possible should provide a more consistent closure rate. This type data is not achievable in an observational study.

As the investigators move into randomized controlled trials, the investigators will maintain these criteria as the investigators strive to develop a predictive healing model when all aspects of patient care are considered. This will include which advanced dressing would be best applied to the wound based on patient status using an Artificial Intelligence program under development.

The investigators will also be looking at historical data on wound closure rates for traditional dressing as well as other advanced dressings that has been collected with similar eligibility criteria. All data input into our model will be controlled by similar eligibility requirements. This data will also be used as historical control for this study.

ELIGIBILITY:
Inclusion Criteria:

* Understands and agrees that the standard treatment protocol will include the application of ProgenaMatrix™ as the standard of care for this project.
* Have participated in the informed consent process and signed a data collection and treatment specific informed consent.
* Be able and willing to comply with the data collection procedures, data collection visits, dressings, and off-loading.
* Have type I or type II diabetes mellitus with an Investigator-confirmed glycosylated hemoglobin (HBA1c) of less than or equal to 11.5% within 3 months prior treatment.
* Have at least one DFU Ulcer that has been in existence for a minimum of 4 weeks but no more than 12 months and meets all the following criteria:

  * Ulcer is partial or full thickness without capsule/tendon/bone exposure.
  * Ulcer is on the foot or ankle.
  * Ulcer area is greater than 1 sq. cm. but less than 18 sq. cm. post debridement. (Ulcers larger than 18 sq. cm. can be included with the approval of the Medical Monitor.)
  * If the subject has more than one ulcer the data collection ulcer will be at the discretion of the Investigator.
  * There is minimum of 1 cm between the ulcer treated and any other ulcer on the same foot.
* Have adequate vascular perfusion of the affected limb as defined by one of the following in order of preference.

  * Ankle-Brachial index of greater than .65 and less the 1.3
  * Toe Pressure of greater than 40 mmHg
  * TcPO2 of greater than 40 mmHg
* Patient had vascular re-perfusion more than 30 days prior to inclusion in the study.

Exclusion Criteria:

* The study ulcer has unexplored tunneling, undermining, or sinus tracts.
* The patient is unable to safely ambulate with appropriate off-loading device.
* The patient has a known sensitivity to the suggested dressings.
* The patient has or is suspected of having gangrene, wound infection, necrosis, redness, pain, purulent drainage or is being treated by antibiotic for the treatment of the above.
* The patient has confirmed osteomyelitis of the foot with the ulcer.
* The patient is on steroid therapy, immunosuppressive or autoimmune therapy, radiation therapy of the foot, thrombosis.
* History of bone of metastatic disease of the affected limb, radiation therapy or chemotherapy within 12 months prior to treatment.
* Pregnancy
* The patient is affected by any disease other than diabetes that can impair wound healing in the opinion of the Investigator.
* The patient has unstable Charcot with bony prominence that will inhibit wound healing.
* Excessive lymphedema that will inhibit off-loading.
* Is unwilling to allow the use ProgenaMatrix™ as the standard of care for this data collection project.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
time to wound closure | 12 weeks of treatment
  The endpoint of this data collection process is to study the timepoint for total wound closure following the protocol procedures in the use of ProgenaMatrix™.

CONTACTS AND LOCATIONS:
Locations (1):
- United Wound Healing, Puyallup, Washington, United States

IPD SHARING:
Plan to Share IPD: No